CLINICAL TRIAL: NCT04216238
Title: Association of Wearable Activity Monitors With Post-Operative Activity Level Among Cardiovascular Surgical Patients
Status: Completed | Type: Observational
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 038.NUR.2019.M
Record Dates: First submitted 2019-08-12; First posted 2020-01-02 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Cardiovascular
Keywords: cardiovascular surgical patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiovascular surgical patients: Patients who received cardiovascular surgery and was released from the hospital due to meeting and exceeding a certain walking distance.
  Interventions: Behavioral: quasi-experimental Pre-test/Post-test design

INTERVENTIONS:
Behavioral: quasi-experimental Pre-test/Post-test design — surveys to document progress

SUMMARY:
Early mobility in the post cardiovascular surgical patient can dramatically impact patient outcomes. Utilizing an innovative strategy, like a wearable activity monitor, can potentially provide: accurate data on post-operative mobility level; increased motivation and self-efficacy in the recovering patient; data to potentially drive post-operative mobility goal setting. Use of a wearable activity monitor will reduce time needed to return to pre-operative activity level in the cardiovascular surgical patient.

DETAILED DESCRIPTION:
While this study used participants from a general surgical floor, its merit should be translatable to the cardiovascular surgical patient population. Additionally, Thorup et al. (2016) proved a positive correlation between the amount of time a step counting device was worn and the distance walked by patients.

It is no surprise that the importance of activity level and ambulation goals are stressed as much, if not more, to cardiac surgery patients versus other surgical patients. In order to be released from the hospital, a cardiac surgery patient must meet and exceed a certain walking distance. Because of this, much of the post-operative teaching is related to the importance of ambulating, setting distance goals, and defining a walking plan to adhere to during the hospital stay and after discharge.

Early and sustained mobility in the post cardiovascular surgical patient can positively impact patient outcomes. In order to drive these outcomes, patient ownership, motivation and self-accountability beyond the walls of the hospital must be achieved.

This study will use best practice guidelines, the relationship-based care model, and innovative technology to determine if using wearable activity monitors impacts: (1) intrinsic motivation, (2) time of return to pre-operative mobility levels, (3) LOS and readmission rates, and (4) overall fitness level.

The aim of this study is to determine if use of a wearable activity monitor will motivate post cardiovascular surgical patients to increase activity levels over a 12 week period, to determine the wearable activity monitor's ability to influence return to pre-surgical self-reported mobility level, to determine if using a wearable activity monitor will increase 6 minute walk test(6MWT) distance comparing pre-discharge 6MWT and 3 month post 6MWT, to determine amicability of a wearable activity monitor as an intervention strategy in post cardiovascular surgical patients, to determine if use of a wearable activity monitor as a post-operative intervention will impact patient length of stay and/or readmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least 18 years old
* Patient must have cardiovascular surgery
* Patient must be able to ambulate without the use of an assistive device
* Patient must be able to wear activity wrist device
* Patient must speak and read English

Exclusion Criteria:

* Patient does not speak or read English
* Patient is not able to ambulate, is wheelchair bound, bed bound, or requires the use of an assistive device for ambulation
* Patient is discharged to an inpatient rehabilitation facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cardiovascular surgical patients will be recruited preoperatively for participation in study with an anticipated three month time commitment. Upon informed consent, participant will receive pre-test and wearable activity monitor hardware from study investigator. The 6 minute walk test will be conducted prior to discharge from the hospital and again during the three month follow-up visit along with the post-test survey.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
intrinsic motivation | over a period of 12 months
  refers to behavior that is driven by internal rewards. In other words, the motivation to engage in a behavior arises from within the individual because it is naturally satisfying.
time of return to pre-operative mobility levels | over a period of 12 months
  time of return to pre-operative mobility levels
LOS | over a period of 12 months
  LENGTH OF STAY
readmission rates | over a period of 12 months
  readmission rates
overall fitness level | over a period of 12 months
  FITNESS LEVEL

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Williams, BSN, RN, Principal Investigator — Methodist Mansfield Medical Center
Locations (1):
- Methodist Mansfield Medical Center, Mansfield, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided